CLINICAL TRIAL: NCT05151731
Title: A Phase II, Multicenter, Randomized, Double Masked, Active Comparator-Controlled Study to Investigate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7200220 Administered Intravitreally in Patients With Diabetic Macular Edema
Brief Title: A Study to Investigate Vamikibart (RO7200220) in Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BP43445; 2021-003756-16 (EudraCT Number)
Record Dates: First submitted 2021-12-08; First posted 2021-12-09 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: 0.25 mg Vamikibart Q8W (Experimental): Participants will receive vamikibart 0.25 milligrams (mg), by intravitreal (IVT) injection, on Day 1 and every 8th week (Q8W), up to Week 44, for a total of 6 injections. A sham procedure will be administered during study visits at which no study drug is administered to maintain masking between treatment arms.
  Interventions: Drug: Vamikibart; Other: Sham Procedure
- Arm B: 1.0 mg Vamikibart Q8W (Experimental): Participants will receive vamikibart 1.0 mg, by IVT injection, on Day 1 and Q8W, up to Week 44, for a total of 6 injections. A sham procedure will be administered during study visits at which no study drug is administered to maintain masking between treatment arms.
  Interventions: Drug: Vamikibart; Other: Sham Procedure
- Arm C: 1.0 mg Vamikibart Q4W (Experimental): Participants will receive vamikibart 1.0 mg, by IVT injection, on Day 1 and every 4th week (Q4W), up to Week 44 for a total of 12 injections.
  Interventions: Drug: Vamikibart
- Arm D: 0.5 mg Ranibizumab Q4W (Active Comparator): Participants will receive ranibizumab 0.5 mg, by IVT injection, on Day 1 and Q4W, up to Week 44 for a total of 12 injections.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Vamikibart — Vamikibart will be administered by IVT injection as specified in each treatment arm.
  Other Names: RO7200220
  Arms: Arm A: 0.25 mg Vamikibart Q8W; Arm B: 1.0 mg Vamikibart Q8W; Arm C: 1.0 mg Vamikibart Q4W
Drug: Ranibizumab — Ranibizumab 0.5 mg will be administered to the participants by IVT injection, as specified in the treatment arm.
  Other Names: Lucentis
  Arms: Arm D: 0.5 mg Ranibizumab Q4W
Other: Sham Procedure — Sham is a procedure that mimics an IVT injection and involves the blunt end of an empty syringe (without a needle) being pressed against the anesthetized eye. Sham procedure will be administered to participants in the Q8W arms at applicable visits to maintain masking between treatment arms.
  Arms: Arm A: 0.25 mg Vamikibart Q8W; Arm B: 1.0 mg Vamikibart Q8W

SUMMARY:
Study BP43445 is a phase II, multicenter, randomized, double-masked, active comparator-controlled study to investigate the efficacy, safety, tolerability, pharmacokinetics, and pharmacodynamics of vamikibart administered intravitreally in participants with diabetic macular edema. Only one eye will be chosen as the study eye. The duration of the study will be up to 76 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus (Type 1 or Type 2)
* Macular thickening secondary to diabetic macular edema (DME) involving the center of the macula
* Decreased visual acuity attributable primarily to DME
* Ability and willingness to provide written informed consent and to comply with the study protocol
* Willingness to allow Aqueous Humor collection
* For women of childbearing potential: agreement to remain abstinent or use at least one highly effective contraceptive method that results in a failure rate of <1% per year during the treatment period and for at least 12 weeks after the final dose of study treatment

Exclusion Criteria:

* Hemoglobin A1c (HbA1c) of greater than (>) 12%
* Uncontrolled blood pressure, defined as a systolic value greater than (>)180 millimeters of mercury (mmHg) and/or a diastolic value >100 mmHg while a patient is at rest
* Currently pregnant or breastfeeding, or intend to become pregnant during the study
* Prior treatment with panretinal photocoagulation or macular laser to the study eye
* Any intraocular or periocular corticosteroid treatment within the past 16 weeks prior to Day 1 to the study eye
* Prior Iluvien or Retisert implants within 3 years prior to Day 1 to the study eye
* Prior or concomitant treatment with anti-VEGF therapy within 8 weeks prior to Day 1 to the study eye; Vabysmo^TM within 16 weeks prior to Day 1, prior Beovu® is not permitted
* Prior administration of IVT brolucizumab (Beovu®): ever; vamikibart: </=24 weeks prior to Day 1) in either eye
* Any proliferative diabetic retinopathy
* Active intraocular or periocular infection or active intraocular inflammation in the study eye
* Any current or history of ocular disease other than DME that may confound assessment of the macula or affect central vision in the study eye
* Any current ocular condition which, in the opinion of the investigator, is currently causing or could be expected to contribute to irreversible vision loss due to a cause other than DME in the study eye
* Other protocol-specified inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) Averaged Over Week 44 and Week 48, in Treatment-naïve Participants | Baseline, Week 44 and Week 48

SECONDARY OUTCOMES:
Number of Participants With Systemic and Ocular Adverse Events (AEs) | Up to Week 72
Number of Participants With Abnormal Laboratory Findings, Abnormal Vital Signs Values, or Abnormal Electrocardiogram (ECG) Parameters | Up to Week 72
Number of Participants With Abnormalities in Standard Ophthalmological Assessments | Up to Week 72
Mean Change From Baseline in BCVA Averaged Over Week 44 and Week 48, in Previously Treated Participants | Baseline, Week 44 and Week 48
Mean Change From Baseline in BCVA Averaged Over Week 44 and Week 48, in Overall Enrolled Population | Baseline, Week 44 and Week 48
Mean Change From Baseline in BCVA Averaged Over Week 20 and Week 24, in Treatment-naïve Participants | Baseline, Week 20 and Week 24
Mean Change From Baseline in BCVA Averaged Over Week 20 and Week 24, in Previously Treated Participants | Baseline, Week 20 and Week 24
Mean Change From Baseline in BCVA Averaged Over Week 20 and Week 24, in Overall Enrolled Population | Baseline, Week 20 and Week 24
Mean Change From Baseline in BCVA Averaged Over Week 32 and Week 36, in Treatment-naïve Participants | Baseline, Week 32 and Week 36
Mean Change From Baseline in BCVA Averaged Over Week 32 and Week 36, in Previously Treated Participants | Baseline, Week 32 and Week 36
Mean Change From Baseline in BCVA Averaged Over Week 32 and Week 36, in Overall Enrolled Population | Baseline, Week 32 and Week 36
Change From Baseline in BCVA Over Time | From baseline up to end of study (up to Week 72)
Percentage of Participants Gaining Greater Than or Equal to (≥) 15, ≥ 10, ≥ 5, or ≥ 0 Letters in BCVA From Baseline Over Time | From baseline up to end of study (up to Week 72)
Percentage of Participants Avoiding a Loss of ≥ 15, ≥ 10, ≥ 5, or ≥ 0 Letters in BCVA From Baseline Over Time | From baseline up to end of study (up to Week 72)
Percentage of Participants With BCVA ≥ 69 Letters (20/40 Snellen Equivalent), or ≥ 84 Letters (20/20 Snellen Equivalent) Over Time | From baseline up to end of study (up to Week 72)
Percentage of Participants With BCVA of Less Than or Equal to (≤) 38 Letters (Snellen Equivalent 20/200) Over Time | From baseline up to end of study (up to Week 72)
Change From Baseline in Central Subfield Thickness (CST) at Week 48 | Baseline, Week 48
Change From Baseline in CST at Week 36 | Baseline, Week 36
Change From Baseline in CST at Week 24 | Baseline, Week 24
Change From Baseline in CST Over Time | From baseline up to end of study (up to Week 72)
Percentage of Participants With Absence of Diabetic Macular Edema (DME) Over Time | From baseline up to end of study (up to Week 72)
Percentage of Participants With Absence of Intraretinal Fluid and/or Subretinal Fluid Over Time | From baseline up to end of study (up to Week 72)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (74):
- United States (36):
  - Win Retina, Arcadia, California
  - Retina Consultants, San Diego, Poway, California
  - Retinal Consultants Med Group, Sacramento, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Colorado Retina Associates, PC, Lakewood, Colorado
  - Emerson Clinical Research Institute LLC, Washington D.C., District of Columbia
  - Rand Eye, Deerfield Beach, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Retina Institute, Orlando, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Retina Specialists of Tampa, Wesley Chapel, Florida
  - Butchertown Clinical Trials, Louisville, Kentucky
  - Cumberland Valley Retina PC, Hagerstown, Maryland
  - Deep Blue Retina PLLC, Southaven, Mississippi
  - Sierra Eye Associates, Reno, Nevada
  - Opthalmic Consultants of LI, Lynbrook, New York
  - University of Rochester Flaum Eye Institute, Rochester, New York
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Meridian Clinical Research, Cincinnati, Ohio
  - Verum Research LLC, Eugene, Oregon
  - EyeHealth Northwest, Portland, Oregon
  - Erie Retinal Surgery, Erie, Pennsylvania
  - Eye Care Specialists, PC, Kingston, Pennsylvania
  - Sewickley Eye Group, Sewickley, Pennsylvania
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Black Hills Eye Institute, Rapid City, South Dakota
  - Retina Consultants of Nashville, Nashville, Tennessee
  - Texas Retina Associates, Arlington, Texas
  - Austin Clinical Research LLC, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Valley Retina Institute P.A., McAllen, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Piedmont Eye Center, Lynchburg, Virginia
  - Wagner Macula & Retina Center, Norfolk, Virginia
- Argentina (9):
  - Organizacion Medica de Investigacion, Buenos Aires
  - Centro Oftalmologico Dr. Charles S.A., Capital Federal
  - Oftalmos, Capital Federal
  - Buenos Aires Mácula, Ciudad Autonoma Buenos Aires
  - Centro Privado de Ojos Romagosa, Córdoba
  - Centro de ojos Loria, Lomas de Zamora
  - Oftar, Mendoza
  - Microcirugía Ocular S.A, Rosario
  - Grupo Laser Vision, Rosario
- Canada (3):
  - Retina Institute of Ottawa, Ottawa, Ontario
  - Toronto Retina Institute, Toronto, Ontario
  - Institut De L'Oeil Des Laurentides, Boisbriand, Quebec
- Czechia (4):
  - Faculty Hospital Ostrava, Ostrava
  - Faculty Hospital Kralovske Vinohrady, Prague
  - General Teaching Hospital Prague, Prague
  - AXON Clinical, Prague
- Poland (7):
  - Niepubliczny Zak?ad Opieki Zdrowotnej PRYZMAT-OKULISTYKA, Gliwice
  - Uniwersyteckie Centrum Kliniczne, Katowice
  - Centrum Medyczne UNO-MED, Krakow
  - SPSK nr 1 w Lublinie, Lublin
  - Centrum Diagnostyki i Mikrochirurgii Oka LENS, Olsztyn
  - LensClinic, Rybnik
  - Caminomed, Tarnowskie Góry
- Emanuelli Research and Development Center LLC, Arecibo, Puerto Rico
- South Korea (5):
  - Yeungnam University Medical Center, Daegu
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Kim's Eye Hospital, Seoul
- Spain (4):
  - Hospital General de Catalunya, Sant Cugat de Valles, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Oftalvist Valencia, Burjassot, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (5):
  - Bristol Eye Hospital, Bristol
  - Gloucestershire Hospitals NHS Foundation Trust, Gloucestershire
  - Royal Surrey County Hospital, Guildford
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Royal Victoria Infirmary, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing